CLINICAL TRIAL: NCT04272021
Title: Multi Neuro-functional Biomarkers for Monitoring the Effects of Treatments in ADHD Children
Acronym: MIMOSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 504
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADHD sample (Experimental): Children with a diagnosis of ADHD
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — standard therapy for ADHD

SUMMARY:
MIMOSA study aims to characterize from behavioral, neurophysiological and neurocognitive perspectives children and adolescents with attention deficit hyperactivity disorder (ADHD), in order to identify a possible biomarker of response to medication treatments. To achieve this aim, in the study children with ADHD (drug naive) are recruited and undergo behavioral and clinical screenings, neurocognitive profile, and neurophysiological evaluation with functional near infrared spectroscopy (fNIRS). ADHD group is evaluated before the beginning of medications, at first dose of medication (only imaging evaluation fNIRS), and after a period of two/three months of continuous treatment with medication.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ADHD according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) criteria;
* drug naive

Exclusion Criteria:

* presence of intellectual disability, neurological diseases, epilepsy, genetic syndromes
* and previous treatment with psychoactive drugs

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
ADHD rating scale | 2-3 months
  Clinical improvement measured with ADHD rating scale, percentage.

SECONDARY OUTCOMES:
CGI-S | 2-3 months
  Clinical improvement measured with CGI-s (Clinical Global Impression - severity)(minimum value: 1 = "normal, not ill"; maximun value: 7 = "very severely ill" )

OTHER OUTCOMES:
Change in functional neuroimaging | 2-3 months
  functional Near Infrared Spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, Italy

IPD SHARING:
Plan to Share IPD: Undecided